CLINICAL TRIAL: NCT07020702
Title: ElectroPhySiological Characterization Of the Arrhythmia Substrate for Sudden Cardiac Death PrEdiction
Acronym: EP-SCOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHUBX 2022/37
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Ventricular Arrhythmia; Cardiomyopathies; Left Ventricular Ejection Fraction Less Then or Equal to 50percent
Keywords: cardiomyopathies; sudden death; Myocardial Infarction
MeSH Terms: conditions — Cardiomyopathies; Death, Sudden; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Implantation of an ICD (Experimental): Patients implanted with an ICD
  Interventions: Device: Implantation of an ICD
- Clinical follow-up (No Intervention): Patients not implanted with an ICD

INTERVENTIONS:
Device: Implantation of an ICD — Implantation of an ICD
  Arms: Implantation of an ICD

SUMMARY:
EP-SCOPE is a prospective, multicentric, non-randomized pilot study that aims to estimate the risk of life-threatening ventricular arrhythmia through use of advanced electrophysiological studies in patients with ischemic or non-ischemic cardiomyopathy with left ventricular ejection fraction (LVEF) <50% and risk factors of ventricular arrhythmia, otherwise not considered for implantation of an implantable cardioverter defibrillator (ICD).

The objective is to assess the effectiveness of a risk stratification strategy based on detailed electrophysiological exploration of the left ventricle and programmed ventricular stimulation.

DETAILED DESCRIPTION:
Responsible for 10% of deaths in the general population, sudden cardiac death is mostly caused by malignant ventricular arrhythmias (80%). These arrhythmias mainly occur in cardiomyopathies (75-90%). Currently, the prevention of sudden death is based on risk stratification according to the evaluation of myocardial contractility with indications for prophylactic ICD implantation reserved for LVEF ≤ 35%. This predictor is notoriously insufficient for several main reasons: 1) While ICDs are indicated in patients with LVEF ≤35%, only a minority (2 -5% per year) will suffer from arrhythmia and therefore benefits from ICD implantation, while all will be subject to potential complications. 2) The majority of sudden death (70-80%) occur in patients with LVEF >35%; while they have a lower arrhythmia risk (1-2% per year), they constitute a population four times larger, which is not stratified. 3) Finally, the cardiomyopathy population is broad, and include distinct clinical scenarios that are not specifically addressed.

While conventional electrophysiological studies only boast a limited number of measurements, the proposed strategy is a detailed electrophysiological characterization of the altered ventricle. Measurements include a detailed mapping of the left ventricle in the basal state and during extrastimuli, and programmed stimulation of the right and left ventricle including the simultaneous recording of the Purkinje system.

Follow-up will be performed for 3 years, looking for the occurrence of major arrhythmic events such as: 1) Appropriate therapy (for VT/VF) delivered by an ICD or 2) documented ventricular arrhythmia on ECG, implantable loop recorder or pacemaker or 3) Clinical sudden death.

ELIGIBILITY:
Inclusion Criteria:

* Patient with cardiomyopathy with 35%<LVEF<50% and at least one risk factor
* Patients with cardiomyopathy with LVEF≤35% and an indication for cardiac resynchronisation

Exclusion Criteria:

* Patients who are minors or aged 80 or over
* Patients with unstable coronary artery disease
* Myocardial infarction less than 40 days old
* Coronary revascularisation <90 days
* Patients with intracardiac thrombus
* Patients with a mechanical heart valve
* Patient implanted with an automatic defibrillator
* Patient life expectancy <1 year
* Pregnant or breast-feeding women
* Anti-arrhythmic drugs other than beta-blockers and amiodarone

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2030-09-12 (Estimated); Study Completion 2030-09-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence of major rhythmic events | 60 months
  Follow-up on Occurrence of major rhythmic events

SECONDARY OUTCOMES:
Surfaces distributions of abnormal ventricular potentials | Day 1
Spatial distributions of abnormal ventricular potentials | Day 1
Purkinje potentials in induced arrhythmias | Day 1
  Presence or absence

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - CHU de Bordeaux - Hôpital Cardiologique du Haut-Lévêque, Pessac
  - CHU de Saint-Etienne, Saint-Etienne